CLINICAL TRIAL: NCT01531543
Title: Phase 4 Study of Primary Use of the Vacuum Assisted Laparostomy in Treatment of Severe Peritonitis
Brief Title: Prospective Comparison of Primary Abdominal Closure and Vacuum Assisted Laparostomy in Treatment of Severe Peritonitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Faculty Hospital Na Bulovce (Other)
Responsible Party: Principal Investigator, Zuzana Serclova, MD, Head of ICU - Department of Surgery, Principal Investigator, The Faculty Hospital Na Bulovce
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BuloVAC
Record Dates: First submitted 2012-02-07; First posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Peritonitis
Keywords: Vacuum Assisted Closure (VAC); Laparostomy; Severe peritonitis
MeSH Terms: conditions — Peritonitis | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAC-laparostomy (Experimental): Primary use of Vacuum Assisted Closure (VAC) laparostomy after surgical revision because of severe peritonitis
  Interventions: Device: V.A.C.- Vacuum assisted closure laparostomy (KCI)
- Primary abdominal closure (No Intervention): The abdominal wall is primary closed after the surgical revision because of severe peritonitis

INTERVENTIONS:
Device: V.A.C.- Vacuum assisted closure laparostomy (KCI) — Primary Vacuum Assisted Closure (V.A.C.)laparostomy was indicated after surgery in patients with severe peritonitis. VAC laparostomy was performed using sandwich technique (semi-permeable foil - intraabdominal foam - dynamic sutura of the fascia - foam inserted subcutaneously - non-permeable foil) and connected to the active suction of 125mmHg.
  Other Names: Vacuum Assisted Closure (V.A.C.) - KCI, USA
  Arms: VAC-laparostomy

SUMMARY:
The aim of the project was to optimalize the process in severe peritonitis which is generally inflicted with high mortality and morbidity with long term costly therapy. Therapy of severe intraabdominal infection consist of treatment of the infection site and following closure of the abdominal cavity with possibility of re-laparotomy and in treatment of complications when needed; or closure introduction of laparostomy with intention to control complications prevention however with risk of tertiary peritonitis. Modern process is laparostomy with active suction (VAC) method which reduces the risk of tertiary peritonitis. It efficacy is however approved especially in therapy of complications. Based on the investigators experiences the investigators use this method even in case of primary treatment of severe peritonitis which led to protocol processing (VAC in case of primary closure of the abdominal cavity; VAC exchange according to scoring system; secondary closure of the abdominal cavity or early coverage with collagen mesh). The aim of this project is to prove reduced mortality, morbidity and hospitalization length (cost reduction) in prospective randomized study in patients treated due to severe peritonitis using VAC method in comparison to classical approach (primary closure of the abdominal cavity; secondary solution of complications).

DETAILED DESCRIPTION:
Introduction Severe peritonitis belongs among severe diseases with mortality 20-60%. Causes are number of primary surgical diseases (inflammatory acute abdomen syndromes - perforated diverticulitis, perforated tumor, colon ischemia and other) or complications after abdominal surgeries in frequency 12-16%.

Secondary and tertiary peritonitis can be in insult causing system inflammatory response (SIRS) with subsequent sepsis and multi-organ failure; it is serious state of patient who requires long term and costly intensive care and despite of that it often ends with permanent disability. Basic therapy of severe peritonitis is surgical treatment of origin of abdominal sepsis, contamination elimination and prevention of postoperative complications. The insufficient capability to manage postoperative complications (polymorbidity, diabetes, inveterate peritonitis, immunosuppressed patient) is often the cause of organ and mutli-organ failure. In case of primary closure of the abdominal cavity and after correct surgical treatment; solution is the early diagnosis of the complications and their urgent sanitation. Mostly from objective reasons there is delay in complication diagnosis and thus adequate treatment. Other negative consequence of primary closure of the abdominal cavity in case of development of intraabdominal complicated healing is the development of intraabaominal hypertension and even compartment syndrome with all negative influences to organ functions. Alternative is to introduce laparostomy which enables simple abdominal cavity control (second look method) using repeated interventions. Classical laparostomy is however continual continuation of the tertiary contamination. According to known literal sources there is no recommendation for means of abdominal cavity closure in the above given surgical disease which is therapeutically more efficient.

One of the modern laparostomy methods is closure of the abdominal cavity using VAC. Method principle is the active suction which is continual and it drains effusion from the abdominal cavity and thus reduces intraabdominal bacterial contamination and also supports blood circulation and vitality of the wound edges. It is a method which fulfills advantages of laparotomy including expansion of the abdominal cavity, effusion drainage quality of which can be controlled; it is a closed system in which there is no risk of external contamination as in case of common laparostomy. Use of VAC method was verified in various wound types with copious secretion (sternotomy, diabetic foot or fascitis). Method of VAC laparostomy was described; however prospective and randomized use in peritonitis has not bee evaluated yet.

Aim of the project: The aim of this project is to prove reduced mortality, morbidity and hospitalization length (cost reduction) in prospective randomized study in patients treated due to severe peritonitis using VAC method in comparison to classical approach (primary closure of the abdominal cavity; secondary solution of complications). Secondary aim is to validate scoring systems and early sepsis markers (cytokines) in algorithm of assessment of severance of severe peritonitis in our conditions and their inclusion in indication for surgical revision. Tertiary aim is to determine group of patient who would profit the most from the method.

Further aim is to compare costs and socio-economic implications of both therapy options.

Hypothesis: Primary introduction for surgical revision due to severe peritonitis reduces postoperative morbidity and mortality in comparison with primary closure of the abdominal cavity.

Indications for repeated intervention improves combination of scoring systems and immunohistochemistry markers.

Methodology

1- assessment of preoperative stave of patient - APACHE II (Acute Physiology and Chronic Health Evaluation, ASA, BMI), severity of clinical and surgical finding.

2 - Assessment of influence of selected method primary treatment of the abdominal cavity on the postoperative morbidity which is expressed by monitoring basic vital functions, SOFA (Sequential Organ Failure Assessment), intraabdominal pressure monitoring, serum level of cytokines monitoring, postoperative complications, surgical revision and length of hospitalization.

3 - long term and socioeconomic consequence (30 days of follow up after discharge - questionnaire, assessment of life quality), cost analysis expended for hospitalization including medication, surgery as well as postoperative outpatient control visits.

Patient with severe peritonitis will be enrolled in study according to Mannheim Peritonitis Index (MPI) - more than 20-25 according to sex; APACHE II more than 10. Expected sample size is total of 50 patients (25 treated using VAC method) versus 25 in control group). Screening will include all patients designer fulfilling SIRS criteria prior abdominal approach and/or displaying symptoms of peritonitis. If patient fulfills these criteria and agrees with inclusion in study, his/her ID is entered in the electronic database which generates inclusion in one out of two groups according randomization scheme - surgery termination using VAC method or primary suture. Excluded patients: young patients younger than 18 years; mental state of patients which does not enable proper information and signature of informed consent form (see bellow) with inclusion in study; further patients who cannot be assume to live longer than 48 hours after surgery (APACHE II, Karnofski, SOFA).

Preoperative care and actual surgical procedure is not the direct subject of study and will be conducted according to so far known procedures. Surgeon will closed the abdominal cavity according randomization at the end of procedure and this fact is in no way affected by actual surgery procedure.

Patient will be treated at the surgical ICU. First exchange of VAC dressing will be conducted after 24-48 hours and subsequently so called on demand (patient health state aggravation defined as score SOFA increase by 4 and more points; elevation of inflammatory markers and interleukins). After complete sanitation of the origin the investigators close the laparostomy (only serous exudate) If it is not technically possible to suture abdominal cavity according to layers, the investigators will close it using following alternatives: single skin cover, mesh plasty, covering with celless skin implant (permacol surgical implant) so the abdominal cavity was closed as soon as possible.

Patient with primary closed abdominal cavity (control group) will be treated according to so far known procedure. In case of inflammation signs the investigators will search and treat this focus. Cytokine inflammatory markers will be also monitored and including finding. In case of surgical complication the investigators will proceed in standard manner (SSI). VAC method will not be used in cases of those patients.

Hospitalization will be terminated after criteria compliance which are: oral intake higher than 2 liters tolerance; sufficient oral analgesics; patient does not display infection signs; agrees with hospitalization; surgical wound is treatable in outpatient clinic.

Means of data collection

Preoperative examination will monitor apart from basic data such as age, diagnosis, co-morbidity score ASA, BMI, level of inflammatory parameters (CRP, blood count, other biochemistry examination). Patient must fulfill criteria SIRS to be enrolled in the study and display signs of peritonitis. Precise indication to surgery will be recorded. After introduction of anesthesia the investigators will perform examination of arterial blood (ASTRUP) and will calculate APACHE

Extent of inflammation (MPI) will be evaluated and source of infection (confirmation or exclusion of preoperative diagnosis). Performed surgical procedure will be described, the investigators will monitor duration of surgery; blood loss; monitoring whether sufficient control of primary source (insufficient treatment of source is sufficient exclusion criterion).

Daily the investigators will monitor IL-1, 6, 8, 10 and TNF alpha while at ICU (during first 5 days), SOFA score will be calculated and IAP will be measured. The investigators will further monitor frequency of VAC exchanges; number of administrated transfusions; duration of UPV; days without oral intake and without possibility of physiotherapy - walking (parameters of recovery. Conscious patients will be submitted form for assessment of life quality (SF-36) on the 7th postoperative day. The investigators will further monitor pain using VAS.

Entry values are: hospitalization length, number of ICU days; mean of wound closure (primary suture, delayed suture after VAC; skin cover and other). Incidence and severity of SSI (I-III grade) and further nosocomial infection (health care - associated infection - HAI). Patient again completes from assessing life quality (SF-36) prior discharge. Active follow up will be in terms of study conducted via telephone every 30th day after discharge. Patient will subsequently complete mailed questionnaire with assessing life quality (SF-36). Outpatient controls will be necessary and repeated hospitalization in complicated patients. After completion of patient monitoring the analysis of cost for hospitalization including medication, surgery and postoperative outpatient control will be conducted using the hospital information system.

Statistical processing

Sample size is estimated based on expected percentage indicator according to Fleisse. Other sample size estimates were estimated using standard method. Each sample must contain 26 -47 patients for mortality estimated between 30-40% and in case of statistically significant difference 20-30% when 5% level of significance and test power 70% in case of one sided test. Morbidity estimated to 60% and clinically significant difference 30-40% requires sample size of 19-32 subjects providing the same significance level and one sided test. Statistical evaluation of results will be included based on pair tests. Difference of individual variables between both groups will be evaluated using Student pair test or its non-parametric variant (Wilcoxon test). SOFA, APACHE II scores and life quality assessment results (SF-36) will be evaluated using Hotelling test as multi directional generalization of Student test.

Time schedule:

1. year of the project: design of randomization program; personal education with study protocol; software design; inclusion of 18 patients. Data processing. Results will be evaluated at the end of the year; statistician will evaluate homogeneity of groups.
2. year of the project: inclusion of further 18 patients. Data analysis will be performed and subgroup analysis and partial results will be processed and presented.
3. year of the project: inclusion of the last 14 patients. Follow up termination. Definite data collection, analysis, results evaluation including financial analysis. Standard proposal. Presentation in national and international forums, publications.

Discussion Surgical treatment is inseparable part of patient care with severe peritonitis. Advance monitoring is important for identification of risk patients but also for possible surgical revision indication. Generally used sepsis markers including scoring systems (APACHE II, MOSF - Multiple Organ System Failure, MODS - Multiple Organ Dysfunction Score) however react with certain delay. Possible or on demand re-laparotomy is performed afterwards in patient in severe conditions with MODS. On the other hand planned re-laparotomies are conducted excessively. Not even met-analysis of clinical studies proved clear preference of one procedure (23). New method VAC however has not been evaluated in prospective randomized study in this indication. Inclusion of early markers of septic state - IL-1, 6, 8, 10 a TNF alpha - in indication for re-laparotomy or VAC exchange could have large clinical benefit. Further controversial indication parameter commonly measured at ICU is size and development of IAP which can present important correlation with laboratory signs of inflammation and it can lead for design of special index. VAC method use has its advantages - active and closed intraabdominal secretion restricts possibilities of spreading HAI. Significant and reduced frequency of dressing; enables simple physiotherapy of patients; condition of anabolic phase which is necessary for any healing (24). Analysis of patient number which benefit from this method (intention-to treat) against general costs is necessary.

Designer's working site has treated 19 patients over the last 18 months using this method. Mortality was 15.8% and average hospitalization length 59.2 days which is in compliance of so far published results. However it has not been prospective randomized study and VAC method was however used as the last therapeutic option.

Information Working site has needed surgical equipment including equipment for performing of VAC; VAC is used as method for 5 years; apart from purchase of consumption material he is the only owner of the pump. This method has been used to treat different wounds. Principal investigator and all co-workers has experience with this method. Co-investigator has even numerous experiences with clinical studies and he published his results in journals. Other specific equipment is not necessary for study procedure.

Conclusion Detected results will background for verification of efficacy of VAC introduction into laparostomy in patients after surgical revision due to severe peritonitis. Efficacy of new and standard laboratory and clinical markers of septic state.

Expected results, aims, priorities and significance of the project Study output will consist of data usable for design of recommended procedure for surgical patient care with severe peritonitis. Standardized protocol will be introduced for ICU patients which reflect only those laboratory methods and clinical parameters which clinically influence therapy. Detailed analysis for both groups will enable precise indication single surgical interventions which will ensure efficient and thus cost wise preferable therapy. Simple universal software will be created in terms of study which manages patient database and thus enables rapid concurrent assessment of health care quality.

With regard that similar complex prospective study has not been published in national and international magazines, publication in impact journal; socioeconomic analysis will be published especially in national medical journals so it would be easily accessible.

ELIGIBILITY:
Inclusion Criteria:

* patients indicated for urgent surgery for suspected acute abdomen with severe peritonitis (meet SIRS criteria or signs of diffuse peritoneal irritation)
* the diagnose of severe peritonitis is confirmed intraoperatively (Mannheim Peritonitis Index - MPI > 25)
* patient agrees with inclusion to the study

Exclusion Criteria:

* patients aged < 18 and > 80 years
* patients with not expected survival longer than 48 hours after surgery
* patients with different peroperative finding
* primary abdominal closure is not technically possible
* pregnant or nursing women
* patient does not agree to participate in the study, self-payers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 60 days after surgery
  The proportion of survivors and died patients

SECONDARY OUTCOMES:
Surgical Site Infection rate | 30 days after surgery
  Incidence of HAIs during the 60 days after surgery. Diagnosis confirmed using criteria CDC/NHSN
Length of stay | duration of hospital stay, an expected average of 3 weeks
  Length of hospital stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Ryska, MD, Principal Investigator — Department of surgical, Faculty Hospital Bulovka, Prague, Czech Republic
Locations (1):
- Faculty Hospital Bulovka, Prague, Czechia